CLINICAL TRIAL: NCT00550732
Title: A Phase II Study on Treatment of Refractory Fungal Infections With Posaconazole. The "TIP" Study.
Brief Title: A Study to Examine the Efficacy and Safety of Posaconazole When Introduced Early in the Treatment of Refractory Fungal Infections (P05090 AM2)
Acronym: TIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: JSS Medical Research Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05090
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2013-12-27 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-03

CONDITIONS: Mycoses
Keywords: Triazoles
MeSH Terms: conditions — Mycoses | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Posaconazole (Experimental): Posaconazole oral suspension was administered as 400 mg twice daily (bis in die, BID) with food or 200 mg four times daily (quater in die, QID) without food for a minimum of 1 month.
  Interventions: Drug: Posaconazole

INTERVENTIONS:
Drug: Posaconazole — Posaconazole oral suspension was administered as 400 mg twice daily (bis in die, BID) with food or 200 mg four times daily (quater in die, QID) without food for a minimum of 1 month.
  Other Names: SCH056592; Noxafil®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of posaconazole in the early treatment of fungal infections in participants who are refractory to, intolerant to, or medically precluded from first-line monotherapy or first-line combination antifungal therapy.

DETAILED DESCRIPTION:
In the past two decades, invasive fungal infections (IFI) have become increasingly common among immunocompromised people, including solid-organ or hematopoietic stem-cell transplant recipients, those with HIV infection, those with hematological malignancies, and individuals on immunosuppressive drug regimens. There is a high rate of morbidity and mortality associated with IFI. Over the past decade, there has been an increase in resistance to commonly used antifungal agents and an epidemiological shift to more drug-resistant strains. This has demonstrated the need for the development of a new generation of azoles.

ELIGIBILITY:
Inclusion Criteria:

* Proven or probable invasive fungal infection (IFI) including breakthrough infection while on antifungal treatment for at least 7 days.
* Refractory or intolerant to prior antifungal therapy, or medically unable to receive standard antifungal therapy.
* Age ≥13 years old.
* Expected to survive >1 month.
* Negative pregnancy test (serum or urine) at baseline for women of childbearing potential.

Exclusion Criteria:

* Serum bilirubin >10 times upper limit of normal (ULN).
* Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >10 times ULN.
* Documented allergy to azoles.
* Unable to take oral suspension medications or enteral feeding.
* Pregnant or breastfeeding.
* Participants who have received an investigational drug are allowed to be enrolled if the investigational drug was given 30 days prior to study registration, unless approved by the Sponsor.
* Requires surgery.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 8 medical centers across Canada.
Period: Overall Study
Arm/Group | Posaconazole
Started | 40
Completed | 29
Not Completed | 11
Not completed — Death | 4
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1
Not completed — Palliative care | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Posaconazole
Number analyzed (Participants) | 40
Age, Customized [Median (Full Range); unit: Years] | 48 [17 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 21

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) by 12 Weeks or End of Treatment
Description: Complete Response was defined as resolution of all attributable clinical signs and symptoms and radiologic and mycologic abnormalities, if present at baseline. Partial Response was defined as clinically meaningful improvement in attributable clinical signs and symptoms and radiologic and mycologic abnormalities, if present at baseline.
Time Frame: Up to 6 months
Population: The Efficacy Population included those participants with both a baseline and at least 1 post-baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 35
Percentage of participants
  Complete Response | 26
  Partial Response | 46

2. Secondary Outcome: Number of Participants With ≥50% Decrease in Lesion Size or Number
Description: Reduction in lesion size was analyzed by computed tomography (CT) scan. An imaging response was defined as >=50% reduction in lesion size for pulmonary and cerebral disease or >=50% reduction in the number of lesions for liver disease.
Time Frame: Up to 6 months
Population: This outcome measure was not reported as the Safety and Steering Committee (SSC) no longer considered it relevant based on revised Mycoses Study Group and European Organization for Research and Treatment of Cancer (MSG/EORTC) Consensus Criteria.
Arm/Group | Posaconazole
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants With a CR or PR by 12 Weeks
Description: as for outcome 1
Time Frame: Up to 12 Weeks
Population: The Efficacy Population included those participants with both a baseline and at least 1 post-baseline assessment.
Measure: Number; unit: Percentage of participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 35
Percentage of participants | 75

4. Secondary Outcome: Percentage of Participants With CR or PR by 4 Weeks and by 26 Weeks
Description: as for outcome 1
Time Frame: Up to 26 weeks
Population: The Efficacy Population included those participants with both a baseline and at least 1 post-baseline assessment.
Measure: Number; unit: Percentage of Participants
Groups:
- Prosaconazole: Posaconazole oral suspension was administered as 400 mg BID with food or 200 mg QID without food for a minimum of one month.
Arm/Group | Prosaconazole
Number analyzed (Participants) | 35
Percentage of Participants
  Week 4, CR | 6
  Week 26, CR | 26
  Week 4, PR | 28
  Week 26, PR | 48

5. Secondary Outcome: Percentage of Participants With Infection-free Survival After the Last Dose of Study Drug
Description: Infection-free survival was the proportion of evaluable participants included in the efficacy analysis who are infection-free and alive at 6 months post last dose visit. Infection-free is defined as the resolution of signs and symptoms of infection.
Time Frame: Up to 6 months
Population: The Efficacy Population included those participants with a visit 6 months after the last dose.
Measure: Number; unit: Percentage of participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 25
Percentage of participants | 56

6. Secondary Outcome: Overall Survival at 3 Months
Description: Total number of participant survivors was assessed at 3 months.
Time Frame: 3 months
Population: All enrolled participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 40
Percentage of Participants | 85

7. Secondary Outcome: Number of Participants With Response to Posaconazole in Combination Therapy
Description: as for outcome 1
Time Frame: Up to 6 months
Population: The proportion of participants with response to posaconzole who received a prior combination antifungal regimen is not reported as per recommendation from the Safety and Steering Committee since only 1 participant was evaluable for this outcome measure.
Arm/Group | Posaconazole
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An adverse event (AE) is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration whether or not considered related to the use of the study drug.
Time Frame: Up to 12 months
Population: All enrolled participants who received at least one dose of study medication.
Measure: Number; unit: Number of participants
Arm/Group | Posaconazole
Number analyzed (Participants) | 40
Number of participants | 39

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: The Safety Population included all enrolled participants who received at least one dose of study medication.
Arm/Group | Posaconazole
Serious Adverse Events (participants affected / at risk) | 16/40
Other Adverse Events (participants affected / at risk) | 35/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=40)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Ludwig angina (Infections and infestations) | 1 (1)
Lung infection pseudomonal (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posaconazole (N=40)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Tachycardia (Cardiac disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 13 (15)
Oral pain (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (6)
Chest pain (General disorders) | 5 (5)
Disease progression (General disorders) | 4 (4)
Fatigue (General disorders) | 7 (7)
Oedema peripheral (General disorders) | 4 (5)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 5 (7)
Bacteraemia (Infections and infestations) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (6)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 8 (8)
Hypoaesthesia (Nervous system disorders) | 4 (6)
Insomnia (Psychiatric disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 6 (6)
Hypotension (Vascular disorders) | 4 (4)
Thrombosis (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigators agree to provide review copies of abstracts or manuscripts for publication (including texts of oral presentations) which report any results of the protocol study to the sponsor, 30 days prior to submission for publication or presentation. The sponsor shall have the right to review and comment on the data analysis and presentation with regard to proprietary information and the accuracy of the information contained in the publication.